CLINICAL TRIAL: NCT00873158
Title: Outcomes Following Dynamic Splinting and/or Physical Therapy for Patients With Adhesive Capsulitis
Brief Title: Dynamic Splinting for Patients With Adhesive Capsulitis
Acronym: DS-SDH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unrelated to trial
Sponsor: Dynasplint Systems, Inc. (Industry)
Collaborators: McMurry University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shoulder 100
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; ROM; Dynasplint
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy Group (No Intervention): Patient's in the Physical Therapy Group will have the standard manual treatments during their usual physical therapy visits with no additional intervention
- Dynasplint Group (Experimental): Along with standard manual physical therapy, patients will have a stretching device (Dynasplint) used in rehabilitation to regain ROM in stiff joints. Patients will use this device 20-30 minutes 2 times per day at home.
  Interventions: Device: Dynasplint

INTERVENTIONS:
Device: Dynasplint — Dynamic splinting utilizes the protocols of Low-Load Prolonged Stretch (LLPS) with calibrated adjustable tension to increase Total End Range Time (TERT)to reduce contracture. The Dynasplint or "Experimental" group will add this therapy to their standard of care regimen
  Arms: Dynasplint Group

SUMMARY:
The purpose of this study is to compare two treatments for adhesive capsulitis.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of two treatment regimens for adhesive capsulitis: dynamic splinting and/or manual physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic adhesive capsulitis
* greater than 50% limitation in active flexion, internal rotation, or external rotation
* Tight GHJ capsule in at least 2 directions
* Capsular end-feel primarily limits ROM
* Age 40- 64
* Normal X-Rays

Exclusion Criteria:

* Acute adhesive capsulitis
* History of Diabetes Mellitus
* Evidence of a cuff tear
* Recent history of trauma
* Evidence of glenohumeral DJD
* History of shoulder surgery
* Calcification of tendonitis demonstrated on a current X-Ray
* Abnormal X-Ray
* Cervical Radiculopathy/brachial plexus lesions
* Less than 2+/5 muscle strength during mid-line manual muscle testing
* Muscle Atrophy
* Presence of associated systematic conditions
* History of prior therapy for current condition
* Manipulation under anesthesia
* Non compliance
* Shoulder-Hand syndrome, Complex Regional Pain Syndrome
* History of prior injections for the current problem
* Patient receiving worker's compensation
* Shoulder symptoms with cervical provocative testing
* Positive X-ray findings in the acromioclavicular or sternoclavicular joints
* Abnormal physical signs or symptoms in the A-C or S-C joint

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Number of physical therapy treatments required | throughout trial
Weeks of Dynasplint treatment | throughout trial

SECONDARY OUTCOMES:
Shoulder Range Of Motion | initial consultation, first visit following injection, and monthly following injection
Sharp FAS Neck and Shoulder | initial consultation, immediatly prior to first treatment following injection, and monthly following injection
Disabilities of Arm, Hand, and Shoulder Questionnaire | initial visit, first visit following injection, and weekly until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Buck Willis, PhD, Study Director — Dynasplint Systems, Inc.
Locations (3):
- United States (3):
  - Gaspar Physical Therapy, Solana Beach, California
  - Andrews Research & Education Institute, Gulf Breeze, Florida
  - University Orthopedics Center, State College, Pennsylvania

REFERENCES:
- [Background] Hamdan TA, Al-Essa KA. Manipulation under anaesthesia for the treatment of frozen shoulder. Int Orthop. 2003;27(2):107-9. doi: 10.1007/s00264-002-0397-6. Epub 2002 Sep 13. PMID 12700935
- [Background] Othman A, Taylor G. Manipulation under anaesthesia for frozen shoulder. Int Orthop. 2002;26(5):268-70. doi: 10.1007/s00264-002-0348-2. Epub 2002 Mar 27. PMID 12378350
- [Background] Placzek JD, Roubal PJ, Freeman DC, Kulig K, Nasser S, Pagett BT. Long-term effectiveness of translational manipulation for adhesive capsulitis. Clin Orthop Relat Res. 1998 Nov;(356):181-91. doi: 10.1097/00003086-199811000-00025. PMID 9917683
- [Background] Omari A, Bunker TD. Open surgical release for frozen shoulder: surgical findings and results of the release. J Shoulder Elbow Surg. 2001 Jul-Aug;10(4):353-7. doi: 10.1067/mse.2001.115986. PMID 11517365
- [Background] Pollock RG, Duralde XA, Flatow EL, Bigliani LU. The use of arthroscopy in the treatment of resistant frozen shoulder. Clin Orthop Relat Res. 1994 Jul;(304):30-6. PMID 8020231
- [Background] Warner JJ, Allen A, Marks PH, Wong P. Arthroscopic release for chronic, refractory adhesive capsulitis of the shoulder. J Bone Joint Surg Am. 1996 Dec;78(12):1808-16. doi: 10.2106/00004623-199612000-00003. PMID 8986657
- [Background] Carette S, Moffet H, Tardif J, Bessette L, Morin F, Fremont P, Bykerk V, Thorne C, Bell M, Bensen W, Blanchette C. Intraarticular corticosteroids, supervised physiotherapy, or a combination of the two in the treatment of adhesive capsulitis of the shoulder: a placebo-controlled trial. Arthritis Rheum. 2003 Mar;48(3):829-38. doi: 10.1002/art.10954. PMID 12632439
- [Background] Arslan S, Celiker R. Comparison of the efficacy of local corticosteroid injection and physical therapy for the treatment of adhesive capsulitis. Rheumatol Int. 2001 Sep;21(1):20-3. doi: 10.1007/s002960100127. PMID 11678298
- [Background] Hannafin JA, Chiaia TA. Adhesive capsulitis. A treatment approach. Clin Orthop Relat Res. 2000 Mar;(372):95-109. PMID 10738419
- [Background] Vermeulen HM, Obermann WR, Burger BJ, Kok GJ, Rozing PM, van Den Ende CH. End-range mobilization techniques in adhesive capsulitis of the shoulder joint: A multiple-subject case report. Phys Ther. 2000 Dec;80(12):1204-13. PMID 11087307
- [Background] Hsu AT, Hedman T, Chang JH, Vo C, Ho L, Ho S, Chang GL. Changes in abduction and rotation range of motion in response to simulated dorsal and ventral translational mobilization of the glenohumeral joint. Phys Ther. 2002 Jun;82(6):544-56. PMID 12036396
- [Background] Hsu AT, Ho L, Ho S, Hedman T. Joint position during anterior-posterior glide mobilization: its effect on glenohumeral abduction range of motion. Arch Phys Med Rehabil. 2000 Feb;81(2):210-4. doi: 10.1016/s0003-9993(00)90143-6. PMID 10668777
- [Background] Hsu AT, Ho L, Ho S, Hedman T. Immediate response of glenohumeral abduction range of motion to a caudally directed translational mobilization: a fresh cadaver simulation. Arch Phys Med Rehabil. 2000 Nov;81(11):1511-6. doi: 10.1053/apmr.2000.9389. PMID 11083357
- [Background] Kirkley A, Griffin S, Dainty K. Scoring systems for the functional assessment of the shoulder. Arthroscopy. 2003 Dec;19(10):1109-20. doi: 10.1016/j.arthro.2003.10.030. PMID 14673454
- [Derived] Gaspar PD, Willis FB. Adhesive capsulitis and dynamic splinting: a controlled, cohort study. BMC Musculoskelet Disord. 2009 Sep 7;10:111. doi: 10.1186/1471-2474-10-111. PMID 19735563